CLINICAL TRIAL: NCT03338062
Title: A Pilot Study to Assess Theragnostically Planned Liver Radiation With Functional DVH Analysis to Optimize Individualized Radiation Therapy
Brief Title: A Pilot Study to Assess Theragnostically Planned Liver Radiation to Optimize Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ryan Rhome,, Assistant Professor- Department of Radiation Oncology, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IUSCC-0604
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Cholangiocarcinoma
Keywords: Radiation Treatment
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Theragnostic SBRT Planning (Experimental): The theragnostic SBRT plan using the HIDA scan was chosen as the plan that reduced the dose of radiation to functional liver without compromising target coverage or tumor control.
  Interventions: Diagnostic Test: Hepatobiliary Iminodiacetic Acid (HIDA) scan
- Standard SBRT Planning (No Intervention): The standard SBRT plan was chosen as the plan that reduced the dose of radiation to functional liver without compromising target coverage or tumor control.

INTERVENTIONS:
Diagnostic Test: Hepatobiliary Iminodiacetic Acid (HIDA) scan — HIDA scan was used as the planning scan for SBRT.
  Arms: Theragnostic SBRT Planning

SUMMARY:
The purpose of this study is to compare radiation treatment plans that are designed for patients with liver cancer. One treatment plan will be created using routine procedures and scans normally performed for radiation treatment planning. The other treatment plan will be created using routine procedures with the addition of two imaging scans; a HIDA (Hepatobiliary Iminodiacetic Acid) scan and an MRI (Magnetic Resonance Imaging) scan. This study will evaluate if adding these imaging scans to treatment planning can reduce the amount of radiation to healthy liver tissue during treatment.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be ≥ 18 years of age at the time of signing informed consent
* Diagnosis of primary liver malignancy (including hepatocellular carcinoma [HCC] or cholangiocarcinoma) or liver metastasis from any primary solid tumor site by characteristic imaging findings on CT or MRI, clinical presentation, and/or pathologic confirmation of diagnosis.
* Subjects with other current or prior malignancies are eligible for this study.
* Patients with liver metastases must have at least one of the following clinical factors that may affect liver function:

  1. History of liver resection (at any time)
  2. History of cirrhosis (any cause), fatty liver disease, or hepatic insufficiency due to any cause
  3. Prior radiation to the upper abdomen including radioembolization
* ECOG (Zubrod) Performance Status 0-2.
* Subjects must have a Child-Turcotte-Pugh (CTP) score ≤ 7 to be eligible.
* Patients who have been previously treated with non-SBRT liver directed therapies may be enrolled on study. At least 3 months must have elapsed between the most recent liver-directed therapy and study entry.
* Ability to provide written informed consent and HIPAA authorization
* Subjects with an allergy to contrast agents may be enrolled at the treating physician's discretion with appropriate pre-treatment and symptom management.

Exclusion Criteria

* Subjects who are pregnant or planning to become pregnant during the study. Women of child bearing potential must have a negative pregnancy test
* Subjects must not have received chemotherapy within 2 weeks of planned 1st day of RT.
* No more than 3 lesions may be treated. The maximum sum of the diameter(s) of the lesion(s) must be ≤6 cm
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (or infections requiring systemic antibiotic treatment), active upper GI ulceration or hemorrhage, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would in the opinion of the investigator limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Rhome, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Started | 10 | 5
Completed | 9 | 5
Not Completed | 1 | 0
Not completed — Alternative Therapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.65) | 64.6 (6.36) | 64.1 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Karnofsky Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Status (KPS) classifies patients based on their functional impairment. Lower KPS = worse survival KPS 100-Normal; no complaints; no evidence of disease KPS 90-Able to carry on normal activity; minor signs/symptoms of disease KPS 80-Normal activity with effort; some signs/symptoms of disease KPS 70-Cares for self; unable to carry on normal activity KPS 60-Requires occasional assistance KPS 50-Requires considerable assistance KPS 40-Disabled; requires special care KPS 30-Severely disabled KPS 20-Very sick; hospitalization necessary KPS 10-Moribund KPS 0-Dead
  Participants
    KPS 100 | 1 | 0 | 1
    KPS 90 | 6 | 3 | 9
    KPS 80 | 3 | 2 | 5
Baseline MELD Score [Mean (Standard Deviation); unit: units on a scale] — Model for end-stage liver disease (MELD) score measures the severity of liver dysfunction. MELD scores range from 6 to 40 and are based on lab tests including serum creatinine, total bilirubin, and INR. The higher the number, the worse the liver function.
  units on a scale | 10.2 (4.8) | 10.8 (3.7) | 10.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Functional Reserve of Liver Between Theragnostic SBRT Planning and Standard SBRT Planning
Description: The functional reserve of the liver for both standard SBRT planning and theragnostic SBRT planning will be calculated for each patient regardless of which plan was ultimately chosen.
  Function reserve of the liver = (number of counts outside 15 Gy isodose line / total number of counts within the liver) * global liver function; where global liver function is the rate of liver uptake (%/min) between 150 to 300 seconds normalized to body surface area (m^2) using the Du Bois method. The difference in functional reserve between the theragnostic plan and the standard plan was calculated for each patient.
Time Frame: Day -1 of Radiation Treatment
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Mean (Standard Deviation); unit: %/min/m^2
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
%/min/m^2 | 0.22 (0.25) | 0.02 (0.07)

2. Secondary Outcome: Percentage of Participants for Whom Theragnostically Planned Radiation is Chosen for the Radiation Treatment Plan
Description: The percentage of participants for whom theragnostically planned radiation is chosen for the radiation treatment plan over the standard plan will be calculated along with the corresponding exact 95% Binomial confidence interval.
Time Frame: Day -1 of Radiation Treatment
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes. The two study arms are combined for this analysis because the arm was assigned based on the SBRT planning scheme that was ultimately chosen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall: All patients who were enrolled on study, received RT, and were assessed for the primary objective.
Arm/Group | Overall
Number analyzed (Participants) | 14
percentage of participants | 64.3 [39.2 to 89.4]

3. Secondary Outcome: Duration of Local Control
Description: Duration of local control was assessed by calculating the time from on study date to date of local failure. Patients who did not experience local failure were censored at their last evaluation date. Local failure (progressive disease at primary diagnosis site) was evaluated using RECIST v1.1 criteria:
  Complete response: Disappearance of all target lesions; Partial response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter; Stable Disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
  The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 15 months
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | NA [NA to NA] — The median and associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data. | NA [3.7 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data.

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from on study date to date of recurrence of any type or death from any cause. Patients who did not experience recurrence or death were censored at their last evaluation date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 15 months
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | NA [1.3 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data. | NA [3.9 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data.

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from on study date to death due to any cause. Patients who remained alive were censored at their last known alive date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 3 years
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | 23.9 [5.2 to 23.9] | 27.5 [1.4 to 27.5]

6. Secondary Outcome: Time to Transplant
Description: Time to transplant was defined as the time from on study date to the date of transplant. Patients who did not receive transplant were censored at their off study date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 15 months
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | NA [NA to NA] — No patients received transplant, so the median and associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data. | NA [NA to NA] — No patients received transplant, so the median and associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data.

7. Secondary Outcome: Time to Distant Liver Failure
Description: Time to distant liver failure was defined as the time from on study date to the date of distant liver failure. Patients who did not experience distant liver failure were censored at their date of last evaluation. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 15 months
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | NA [3.8 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data. | NA [3.9 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data.

8. Secondary Outcome: Time Until Salvage Treatment
Description: Time until salvage treatment was defined as the time from on study date to the start date of salvage treatment. Patients who did not receive salvage treatment were censored at their off study date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 15 months
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
months | NA [2.5 to NA] — The median and one of the associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data. | NA [NA to NA] — The median and associated confidence intervals were not estimable. The median was not reached and the Kaplan-Meier estimate makes no inference about survival times beyond the range of times found in the data.

9. Secondary Outcome: Number of Patients With Treatment-Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event with grade 3 or greater using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Every 15 days for approximately 6 months
Population: Patients who received at least one dose of radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
Participants | 0 | 0

10. Secondary Outcome: Change in MELD Score
Description: Model for end-stage liver disease (MELD) score measures the severity of liver dysfunction. MELD scores range from 6 to 40 and are based on lab tests including serum creatinine, total bilirubin, and INR. The higher the number, the worse the liver function.
Time Frame: Up to 1 year
Population: Patients who received at least one dose of radiation and completed both SBRT planning schemes. Patient numbers differ due to missed visits and/or patients no longer being on study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline MELD Score | 8.8 (1.9) | 10.8 (3.7)
  Change from Baseline to Mid-Treatment: number analyzed (Participants) | 8 | 5
  Change from Baseline to Mid-Treatment | 0.4 (1.7) | -0.4 (0.5)
  Change from Baseline to 1 Month | 0.2 (1.2) | 1.8 (8.6)
  Change from Baseline to 3 Month: number analyzed (Participants) | 9 | 4
  Change from Baseline to 3 Month | 0.8 (3.9) | -2.0 (2.8)
  Change from Baseline to 6 Month: number analyzed (Participants) | 8 | 4
  Change from Baseline to 6 Month | 1.0 (1.9) | -2.0 (3.7)
  Change from Baseline 12 Month: number analyzed (Participants) | 7 | 4
  Change from Baseline 12 Month | 1.4 (1.8) | -1.8 (2.1)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Theragnostic SBRT Planning | Standard SBRT Planning
All-Cause Mortality (participants affected / at risk) | 4/9 | 2/5
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/5
Other Adverse Events (participants affected / at risk) | 9/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theragnostic SBRT Planning (N=9) | Standard SBRT Planning (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theragnostic SBRT Planning (N=9) | Standard SBRT Planning (N=5)
Anemia (Blood and lymphatic system disorders) | 5 (12) | 2 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (3) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (4) | 2 (2)
INR increased (Investigations) | 2 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (7) | 4 (7)
Platelet count decreased (Investigations) | 2 (4) | 3 (5)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT03338062/Prot_SAP_001.pdf
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03338062/ICF_003.pdf